CLINICAL TRIAL: NCT06255847
Title: A Multicenter, Open-label Clinical Study of a Reduced-dose Pomalidomide and Cyclophosphamide Combined With Dexamethasone Regimen for the Treatment of Patients With Debilitating Relapsed-refractory Multiple Myeloma
Brief Title: Clinical Study of Reduced-dose Pomalidomide and Cyclophosphamide Combined With Dexamethasone in the Treatment of Patients With Debilitating RRMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-2022-073
Record Dates: First submitted 2024-01-15; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma in Relapse
MeSH Terms: interventions — pomalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reduced-dose pomalidomide/cyclophosphamide/dexamethasone (PCd) regimen group (Experimental)
  Interventions: Drug: Pomalidomide, cyclophosphamide combined with dexametha

INTERVENTIONS:
Drug: Pomalidomide, cyclophosphamide combined with dexametha — The starting dose of pomalidomide was 2 mg in all cases，the starting dose of cyclophosphamide was 50 mg/day.If the adverse event is attributable to a specific study drug, the dose is reduced accordingly for that drug; if the adverse event is associated with multiple drugs, the dose is reduced appropriately for one of the predominantly associated drugs at the discretion of the investigator; and if multiple adverse events occur concurrently, the dose should be adjusted according to the guidelines for the most severe toxicity.

SUMMARY:
This is an open-label clinical study to evaluate the efficacy and safety of a multicenter, open-label clinical study of a base-reduced-dose pomalidomide, cyclophosphamide combined with dexamethasone (PCd) regimen for the treatment of patients with debilitating relapsed refractory multiple myeloma.

Subjects meeting the enrollment criteria were screened for entry into the study and treated with the appropriate regimen; all patients enrolled in the study did not receive medications other than those specified in the regimen for the treatment of myeloma during the study period, except for supportive care. The primary endpoint of the study is ORR; secondary study endpoints include efficacy above VGPR, progression-free survival (PFS), overall survival (OS), TTNT, safety, and life scale assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with relapsed/refractory MM, including extramedullary infiltration (meeting IMWG 2016 diagnostic criteria);
* IMWG frailty assessment: frail patients.
* Patients with multiple myeloma who have relapsed after previous treatment with 1-3 regimens;
* Patients unresponsive or unable to undergo autologous stem cell transplantation and with disease progression or resistance after prior treatment with proteasome-containing inhibitors (bortezomib) or immunomodulators (thalidomide, lenalidomide); tolerant to more than one of the above drugs;
* Serum monoclonal protein (M protein) reaches measurable levels: serum M protein ≥ 5 g/L; or 24h urinary light chain > 200mg; or serum free light chain > 10mg/dL;
* The patient's clinical indicators must meet the following criteria:ANC ≥ 1.0 x 109/L and PLT ≥ 75 x 109/L for myeloma cells < 50%; any ANC and PLT ≥ 50 x 109 for myeloma cells ≥ 50%; platelets or granulocyte colony-stimulating factor (G-CSF) may be infused to help patients meet the eligibility criteria, but are not permitted within the first 3 days of enrollment; Patients with a glomerular filtration rate ≥10 mL/min who do not require dialysis;
* Patients who have not undergone major surgery, radiation therapy, or participated in another research trial within 2 weeks and have recovered from clinical toxicity of prior therapy;
* with follow-up conditions. Patients understand the characteristics of the disease they suffer from and voluntarily enroll in this study protocol for treatment and follow-up;
* Informed consent has been signed. Informed consent was signed by the patient himself/herself or his/her immediate family members. From the patient's condition, if the patient's own signature is not conducive to the treatment of the condition, then the legal guardian or the patient's immediate family members will sign the informed consent.

Exclusion Criteria:

* Patients with newly diagnosed multiple myeloma (NDMM), plasma cell leukemia;
* Previous use of pomalidomide, cyclophosphamide;
* patients with cyclophosphamide, dexamethasone allergy/intolerance;
* patients with active hepatitis B (HBV), hepatitis C (HCV), and other acquired and congenital immunodeficiency diseases;
* hepatic insufficiency (bilirubin > 3.1mg/100m, ALT and AST > 2 times the upper limit of normal value);
* The presence of severe thrombotic events before treatment;
* Patients with comorbid uncontrolled or severe cardiovascular disease, including myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) defined class III-IV heart failure, uncontrolled angina, clinically significant pericardial disease or cardiac amyloidosis;
* Infection requiring systemic antibiotic therapy, or other serious infection within 14 days;
* Those who underwent major surgery within 30 days prior to enrollment;
* those who require medication for epilepsy, dementia and other abnormal mental conditions who are unable to understand or comply with the study protocol;
* Patients with serious physical or mental illnesses that, in the judgment of the protocol or the investigator, are likely to interfere with participation in this clinical study;
* Substance abuse, medical, psychological, or social conditions that may interfere with the subject's participation in the study or the evaluation of study results;
* persons who, in the opinion of the investigator, are not suitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 12 months
  Overall Response Rate

SECONDARY OUTCOMES:
Efficacy above VGPR | up 3 years
  Stringent complete response is defined as fulfilling the criteria for CR combined with a normal serum free light chain ratio and the absence of clonal plasma cells in the bone marrow as confirmed by immunohistochemistry.
  CR is negative serum and urine immunofixation electrophoresis, disappearance of soft tissue plasmacytomas, and <5% plasma cells in the bone marrow.
  Very good partial response (VPR) is a serum protein electrophoresis with no detectable M protein, but serum and urine immunofixation electrophoresis are still positive; or a reduction in M protein of ≥90% and urinary M protein <100mg/24h.
PFS | within 2 years
  progression-free survival (within 2 years)
OS | up to 2 years
  overall survival
duration from start of study treatment with all 3 agents to start of any new line of treatment | up to 3 years
safety of drugs | up to 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 and EORTC QLQ-C30.
life scale assessment above VGPR（very good partial response） | up to 3 years
  EORTC QLQ-C30 (1-3 months/dose)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomin Zhang, Principal Investigator — Shanxi Bethune Hospital
Locations (1):
- ShanxiBethuneH, Taiyuan, Shanxi, China